CLINICAL TRIAL: NCT06940414
Title: Prevalence and Risk Factors of Hyperkalemia in Non-Dialysis Chronic Kidney Disease Patients in a Community-Based Primary Care Setting
Brief Title: Prevalence and Risk Factors of Hyperkalemia in Non-Dialysis Chronic Kidney Disease Patients in Community
Status: Recruiting | Type: Observational
Sponsor: Xiujuan Zang (Other Government)
Responsible Party: Sponsor-Investigator, Xiujuan Zang, Chief of Nephrology, Songjiang Hospital Affiliated to Shanghai Jiaotong University School of Medicine
Organization: Songjiang Hospital Affiliated to Shanghai Jiaotong University School of Medicine (Other Government)
Other Study IDs: 2025-55-SJ-IRB
Record Dates: First submitted 2025-04-11; First posted 2025-04-23 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-04

CONDITIONS: Hyperkalemia; Chronic Kidney Disease(CKD)
Keywords: Hyperkalemia; Chronic Kidney Disease; Community-Based; Non-Dialysis; Prevalence; Eaglenos POCT System
MeSH Terms: conditions — Hyperkalemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — This is an observational study with no interventions. POCT devices, provided by Eaglenos Sciences, Inc., are used to measure blood glucose, creatinine, uric acid, hemoglobin, and potassium levels in non-dialysis CKD patients for data collection purposes only.

SUMMARY:
The goal of this observational study is to investigate the prevalence and risk factors of hyperkalemia in community-based non-dialysis chronic kidney disease (CKD) patients. The main questions it aims to answer are:

1. What is the prevalence of hyperkalemia in non-dialysis CKD patients in a primary care setting?
2. What are the key risk factors influencing the occurrence of hyperkalemia in this population? Researchers will collect clinical and demographic data from participants across 18 community health centers and use both point-of-care testing (POCT) and laboratory-based methods to measure serum potassium levels and related parameters.

Participants will:

1. Provide blood samples for POCT and laboratory testing.
2. Participate in interviews or questionnaires to gather clinical and lifestyle information.

The findings will be used to construct a risk prediction model for hyperkalemia, aiming to optimize screening pathways and improve disease management strategies in primary care.

DETAILED DESCRIPTION:
Hyperkalemia is a common and life-threatening complication in CKD, with limited data available for non-dialysis patients in community settings. This cross-sectional study will enroll 2,000 non-dialysis CKD patients (Stages 1-5) from 18 community health centers in Songjiang, Shanghai.

The study includes:

1. Validation phase: 500 participants to validate POCT devices for measuring whole blood potassium, glucose, creatinine, uric acid, and hemoglobin.
2. Main phase: 1,500 participants to assess hyperkalemia prevalence and risk factors.

Data will be collected through:

1. POCT and laboratory testing of blood samples.
2. Structured questionnaires capturing demographics, comorbidities, and lifestyle factors.

Statistical analyses will identify key risk factors, and a predictive model will be developed to guide early screening and intervention. This study aims to improve CKD management in primary care by providing evidence for targeted hyperkalemia screening and prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older with stable vital signs, specifically defined as:

  1. Body temperature: 36.0°C-38.0°C;
  2. Pulse: 50-120 beats/min;
  3. Respiratory rate: 10-24 breaths/min;
  4. Blood pressure: Systolic blood pressure ≥90 mmHg and diastolic blood pressure ≥60 mmHg.
* Willing to participate in the study and sign the informed consent form.
* Hematocrit (Hct) level between 25% and 60%.
* Confirmed diagnosis of chronic kidney disease (CKD).

Exclusion Criteria:

* Patients in the unstable phase of acute cardiovascular or cerebrovascular diseases (e.g., acute cerebral infarction, cerebral hemorrhage, or acute coronary syndrome).
* Patients in the unstable phase of severe acute diabetic complications (e.g., diabetic ketoacidosis or hyperosmolar hyperglycemic coma).
* Patients currently in the acute kidney injury (AKI) stage.
* Patients who have started renal replacement therapy.
* Pregnant or breastfeeding women.
* Patients currently participating in or who have participated in other clinical trials within the past six months.
* Patients unable to understand verbal or written instructions, including informed consent content.
* Patients unable to cooperate with the study procedures.
* Other conditions deemed unsuitable for participation in this clinical trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-dialysis CKD patients (Stage 1-5), aged 18 years or older, recruited from 18 community health centers in Songjiang District, Shanghai.
Sampling Method: Non-Probability Sample
Enrollment: 1890 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Hyperkalemia. | At the time of enrollment
  The proportion of non-dialysis CKD patients with hyperkalemia, defined as a blood potassium level greater than 5.0 mmol/L, measured using point-of-care testing (POCT) at enrollment.

SECONDARY OUTCOMES:
Association Between Hyperkalemia and Age. | At the time of enrollment
  Evaluates the association between hyperkalemia (blood potassium > 5.0 mmol/L) and age (years) in non-dialysis CKD patients at enrollment, reported as odds ratios from univariate and multivariate logistic regression analyses.
Association Between Hyperkalemia and CKD Stage. | At the time of enrollment
  Evaluates the association between hyperkalemia (blood potassium > 5.0 mmol/L) and CKD stage (1-5) in non-dialysis CKD patients at enrollment, reported as odds ratios from univariate and multivariate logistic regression analyses.
Association Between Hyperkalemia and Blood Glucose. | At the time of enrollment
  Evaluates the association between hyperkalemia (blood potassium > 5.0 mmol/L) and blood glucose (mmol/L) in non-dialysis CKD patients using POCT at enrollment, reported as odds ratios from univariate and multivariate logistic regression analyses.
Association Between Hyperkalemia and Creatinine. | At the time of enrollment
  Evaluates the association between hyperkalemia (blood potassium > 5.0 mmol/L) and creatinine (μmol/L) in non-dialysis CKD patients using POCT at enrollment, reported as odds ratios from univariate and multivariate logistic regression analyses
Association Between Hyperkalemia and Uric Acid. | At the time of enrollment
  Evaluates the association between hyperkalemia (blood potassium > 5.0 mmol/L) and uric acid (μmol/L) in non-dialysis CKD patients using POCT at enrollment, reported as odds ratios from univariate and multivariate logistic regression analyses.
Association Between Hyperkalemia and Hemoglobin. | At the time of enrollment
  Evaluates the association between hyperkalemia (blood potassium > 5.0 mmol/L) and hemoglobin (g/L) in non-dialysis CKD patients using POCT at enrollment, reported as odds ratios from univariate and multivariate logistic regression analyses.
Performance of Hyperkalemia Prediction Model. | At the time of enrollment
  Assesses the performance of a hyperkalemia prediction model in non-dialysis CKD patients using data from enrollment, reported as area under the ROC curve (AUC), sensitivity (%), and specificity (%).

CONTACTS AND LOCATIONS:
Overall Officials: Xiujuan Zang, MD, Principal Investigator — Songjiang Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Songjiang Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: Data will be made available to qualified researchers upon submission of a research proposal and executionof a data use agreement. Data access will be granted after the final study results are published and after anethical review by the institution's ethics board. Data sharing will be coordinated via email. Qualifiedresearchers can contact zxyykjb@163.com to request access to the data.

REFERENCES:
- [Background] Sevamontree C, Jintajirapan S, Phakdeekitcharoen P, Phakdeekitcharoen B. The Prevalence and Risk Factors of Hyperkalemia in the Outpatient Setting. Int J Nephrol. 2024 Jan 22;2024:5694131. doi: 10.1155/2024/5694131. eCollection 2024. PMID 38292832
- [Background] Sinnathamby ES, Banh KT, Barham WT, Hernandez TD, De Witt AJ, Wenger DM, Klapper VG, McGregor D, Paladini A, Ahmadzadeh S, Shekoohi S, Kaye AD, Varrassi G. Hyperkalemia: Pharmacotherapies and Clinical Considerations. Cureus. 2024 Jan 26;16(1):e52994. doi: 10.7759/cureus.52994. eCollection 2024 Jan. PMID 38406030
- [Background] Einhorn LM, Zhan M, Hsu VD, Walker LD, Moen MF, Seliger SL, Weir MR, Fink JC. The frequency of hyperkalemia and its significance in chronic kidney disease. Arch Intern Med. 2009 Jun 22;169(12):1156-62. doi: 10.1001/archinternmed.2009.132. PMID 19546417
- [Background] Gilligan S, Raphael KL. Hyperkalemia and Hypokalemia in CKD: Prevalence, Risk Factors, and Clinical Outcomes. Adv Chronic Kidney Dis. 2017 Sep;24(5):315-318. doi: 10.1053/j.ackd.2017.06.004. PMID 29031358
- [Background] De Nicola L, Di Lullo L, Paoletti E, Cupisti A, Bianchi S. Chronic hyperkalemia in non-dialysis CKD: controversial issues in nephrology practice. J Nephrol. 2018 Oct;31(5):653-664. doi: 10.1007/s40620-018-0502-6. Epub 2018 Jun 7. PMID 29882199
- [Background] Montford JR, Linas S. How Dangerous Is Hyperkalemia? J Am Soc Nephrol. 2017 Nov;28(11):3155-3165. doi: 10.1681/ASN.2016121344. Epub 2017 Aug 4. PMID 28778861
- [Background] Zhang L, Wang F, Wang L, Wang W, Liu B, Liu J, Chen M, He Q, Liao Y, Yu X, Chen N, Zhang JE, Hu Z, Liu F, Hong D, Ma L, Liu H, Zhou X, Chen J, Pan L, Chen W, Wang W, Li X, Wang H. Prevalence of chronic kidney disease in China: a cross-sectional survey. Lancet. 2012 Mar 3;379(9818):815-22. doi: 10.1016/S0140-6736(12)60033-6. PMID 22386035
- [Background] Ene-Iordache B, Perico N, Bikbov B, Carminati S, Remuzzi A, Perna A, Islam N, Bravo RF, Aleckovic-Halilovic M, Zou H, Zhang L, Gouda Z, Tchokhonelidze I, Abraham G, Mahdavi-Mazdeh M, Gallieni M, Codreanu I, Togtokh A, Sharma SK, Koirala P, Uprety S, Ulasi I, Remuzzi G. Chronic kidney disease and cardiovascular risk in six regions of the world (ISN-KDDC): a cross-sectional study. Lancet Glob Health. 2016 May;4(5):e307-19. doi: 10.1016/S2214-109X(16)00071-1. PMID 27102194